CLINICAL TRIAL: NCT05837962
Title: Feasibility and Acceptability of the Nursing Intervention "EducaTHE" to Improve Knowledge and Self-care Behaviors in the Face of Hypertensive Disorders of Pregnancy in Pregnant Women.
Brief Title: Nursing Intervention for Knowledge and Self-care Behaviors in the Face of Hypertensive Disorders of Pregnancy
Acronym: EducaTHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Edier Mauricio Arias Rojas, Profesor Facultad de Enfermería, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Acta No 234 CEI-FE
Record Dates: First submitted 2023-04-02; First posted 2023-05-01 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Hypertensive Disorders of Pregnancy
Keywords: Knowledge,Self Care,Pregnancy,Nursing, Feasibility Studies

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nursing intervention to improve knowledge and self-care behaviors in the face of HDP (Experimental): Behavioral: Educational, behavioral and motivational intervention developed by nurses aimed at improving the level of knowledge and self-care behaviors of pregnant women in the face of HDP.
  Interventions: Behavioral: Nursing intervention to improve knowledge and self-care behaviors in the face of HDP
- Usual management during prenatal care (No Intervention): Behavioral: Nursing education about maternal care and usual education in maternity preparation course

INTERVENTIONS:
Behavioral: Nursing intervention to improve knowledge and self-care behaviors in the face of HDP — The nursing professional will perform 1 session weekly, for 4 weeks, lasting 90 minutes each. The contents that make up each of the sessions are:
  Session 1. Knowledge about the risk factors, signs and symptoms, maternal and fetal complications of HDP.
  Session 2. Control over behaviour, positive attitude and family and social support: essential components for conducting self-care behaviour.
  Session 3. Nutritional recommendations: eating healthy helps prevent or reduce the risk of developing HDP.
  Recommendations to improve sleep, rest and physical exercise: key routines in my health to prevent or reduce the risk of developing HDP.
  Session 4. Mental health promotion: managing my stress, anxiety and depression levels help prevent or decrease the risk of HDP
  Arms: Nursing intervention to improve knowledge and self-care behaviors in the face of HDP

SUMMARY:
Hypertensive disorders of pregnancy (HDP) are a leading cause of maternal and fetal morbidity and mortality worldwide. The lack of knowledge and self-care behaviors by the pregnant woman in the face of THE could be associated with their appearance. This is a randomized controlled pilot trial type study, with a control group that will receive the usual prenatal care and an intervention group that will additionally receive the nursing intervention to improve knowledge and self-care behaviors in the face of HDP. Each group will include 30 pregnant women, for a total of 60 users. The level of knowledge and self-care behaviors will be assessed before and after the intervention.

DETAILED DESCRIPTION:
Introduction: the World Health Organization (WHO) indicates that HDP are the third leading cause of maternal death worldwide; and in Latin America and the Caribbean they are positioned as the first cause. The evidence has described that limited or non-existent knowledge and the lack of self-care behaviors by the pregnant woman in the face of HDP are important conditions in the incidence of this obstetric complication. In this sense, nursing must design and implement intervention strategies that have a positive impact on knowledge and self-care behaviors in the face of HDP.

Objective: to determine the feasibility and acceptability of the "EducaTHE" nursing intervention to improve knowledge and self-care behaviors in the face of hypertensive disorders of pregnancy in pregnant women.

Methods: randomized controlled pilot trial experimental study with pregnant women assigned to an intervention group and a control group. The sample will consist of a total of 40 pregnant women, 20 in each of the study groups.

The intervention group will receive the usual education of prenatal control. The control group, in addition to the usual prenatal control information, will receive an educational, behavioral and motivational intervention related to HDP and their self-care behaviors. The intervention will be carried out in 4 sessions, on a weekly basis, in a face-to-face and group. In both groups, knowledge and self-care behaviors will be measured before and 4 weeks after the end of the intervention.

Randomization: the assignment will be carried out through a simple randomization process, with an intervention/control ratio 1:1, by means of a sequence of random numbers generated by a statistical program. The assignment will be given by one of the researchers who will not perform the intervention, nor the initial or final evaluation.

Expected results: feasibility and acceptability of the study in the context of perinatal maternal care

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women enrolled in the prenatal care program of a health institution
* Pregnant women aged 18 years or older
* Pregnant women with a gestational age equal to or less than 24 weeks determined by the date of the last period or obstetric ultrasound.
* Pregnant women residing in the urban area.

Exclusion Criteria:

* Pregnant women with chronic conditions such as heart disease, renal disease, or diabetes mellitus.
* Pregnant women with a history or diagnosis at entry or during the study of HDP according to the classification of the American College of Obstetricians and Gynecologists (ACOG)
* Pregnant women who are participating in other educational studies or workshops/programs with similar themes to this study.
* Pregnant women scoring less than 24 points on the Mini-mental status test.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Feasibility: recruitment, attrition, follow-up | 6 months
  Recruitment For the analysis of this variable, the number of pregnant women enrolled in the prenatal control program of the health institution who meet the inclusion criteria of the study, and the number of pregnant women who agree to participate in the study, will be taken into account.
  Attrition This variable will include the number of pregnant women who agreed to participate, and the number of participants who did not attend or did not complete the four sessions of the intervention.
  Follow-up This variable will include the number of pregnant women who complete the four sessions of the intervention, and the number of participants who completed the study after the post-intervention measurements.
Acceptability | 6 months
  A survey will be used to assess acceptability. The survey will be divided into three sessions, the first consisting of 13 items aimed at obtaining information related to the contents of the educational material, the activities and the form of delivery of the intervention, dose and interventionist. The second session consisted of 11 items that will evaluate the benefits and weaknesses of the intervention. The third contains 3 open questions related to the taste for the intervention, suggestions and recommendations

CONTACTS AND LOCATIONS:
Overall Officials: Edier Arias Rojas, Study Director — Universidad de Antioquia; Iliana Ulloa Sabogal, Principal Investigator — Universidad de Antioquia
Locations (1):
- Local Hospital of Piedecuesta, Santander, Piedecuesta, Colombia